CLINICAL TRIAL: NCT03104348
Title: Screening for COPD in Primary Care: a Synergistic Approach - Dentists - Pharmacists -Physiotherapists - Nurses - Physicians
Acronym: UNANIME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very important delay in the pace of inclusions. Likely overestimation of the potential for inclusion. Lack of involvement of some health professionals.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC17.0022 UNANIME
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: COPD
Keywords: COPD; Primary care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD screening (Other)
  Interventions: Diagnostic Test: COPD screening

INTERVENTIONS:
Diagnostic Test: COPD screening — Self-questionnaire with 5 questions Fagerström's test Spirometry

SUMMARY:
A recent French study conducted in the general population in the north, using more than 12,000 people randomly drawn from the electoral lists, shows a prevalence of nearly 15% of an obstructive spirometric function disorder; The diagnosis was ignored in 70% of cases. If we consider the Finistère situation, the mortality data are unfavorable, with an excess of COPD mortality compared to the French average.

Compared to other frequent chronic conditions, such as high blood pressure or diabetes, the management of COPD may appear complex for at least two reasons:

* Screening is difficult because of the banality of symptoms and the need for spirometry to confirm the diagnosis;
* Comorbidities are masking the respiratory pathology; It is on this first point concerning the difficulty of screening that this project focuses.

It is true that the development of screening strategies for COPD has been the subject of numerous studies, the results of which are controversial. The target population of smokers over the age of 40, who are readily selected, is difficult to achieve as a whole because the use of care is far from homogeneous. Many people do not have a general practitioner.

Recent reviews of COPD screening do not recommend systematic screening for COPD in adults. However, they emphasize the feasibility of screening by questionnaire and / or portable spirometry. A selection of patients suspected of exacerbations (patients with at least one episode labeled "bronchitis") could increase the cost-effectiveness of screening by focusing on the most severe cases.

In France, the High Authority for Health (HAS), inspired by the work of the WHO (GOLD programs), offers a simple five-question questionnaire available online for all healthcare professionals in order to facilitate an indication of screening spirometry, where the proposed approach combines symptom identification with active smoking. General practitioners are in this first line of approach for the diagnosis: in fact, the HAS, in its guide of the "pathway of care of the patient COPD", recommends that the general practitioner can carry out the spirometric screening. The corresponding pulmonologist intervenes in this course by completing the explorations and optimizing the management, especially in patients with frequent exacerbations. This ideal scheme is hampered by the present practical organization, a minority of general practitioners (10%) practicing in multidisciplinary health centers, places where the organization of a functional respiratory measurement can be easier.

The current recommendations for smoking cessation allow the coding of this management. It is global, applicable in primary care. It proposes as a starting point the minimal advice, then associates medicines of assistance with the stop, cognitive-behavioral therapies and a prolonged follow-up of the patients after weaning. However, although these comprehensive management techniques are effective for smoking cessation, it is shown that they are underutilized in routine practice by health professionals with low patient participation rates. This is noticed, whereas the application of the minimum board alone would allow about 200 000 people to have access to weaning every year.

In a complementary way, the performance of a functional respiratory test in the active smoking patient has been proposed as a full-fledged tool for the weaning assistance process. Analysis of the literature, however, yields discordant results. Two recent studies have revived the debate: they highlight the potential of spirometry as a communication medium in the context of smoking cessation (using pulmonary age) by confronting patients with the discovery and understanding of their ventilatory disorder obstructive.

Finally, if other health care providers are invited to participate actively in screening, including pharmacists, their place in this screening strategy has been less valued. In particular, pharmacists and dentists are required to provide care to patients with little or no use of the general practitioner: screening for COPD among these patients deserves consideration. Similarly, nurses occupy a special place, being called in particular to carry out regular care of patients, both in their office and at home. The administration of injectable antibiotics in a context of exacerbation of unlikely COPD is a frequent care opportunity, which may include this more comprehensive approach. Finally, physiotherapists, who are increasingly trained in the concept of respiratory rehabilitation, are taking charge of other potentially COPD smokers for other pathologies.

Based on the willingness of Finnish actors to work on a COPD pathway with the help of the regional health agency, the investigators propose to question the respective place of health care professionals involved in primary care among potentially COPD patients: Dentists, nurses, general practitioners, physiotherapists and pharmacists

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years,
* Smoking greater than 10 packs / year, active.
* No previous diagnosis of COPD
* Signature of informed consent

Exclusion Criteria:

* Patients under 40 years of age
* Previous of COPD diagnosis
* Refusing to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness of a COPD screening procedure on primary care with a questionnaire and a measure with a micro-spirometer | 2 months
  Evaluate the effectiveness of a COPD screening procedure in primary care with a questionnaire and an estimate of the FEV1 / FVC ratio by a micro-spirometer, in primary gare

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Charles Yannick, Brest
  - Morvan Pierre-Yves, Brest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hourmant B, Gobert CG, Plumet R, Lott MC, Zabbe C, Tromeur C, Leroyer C, Couturaud F. Screening for COPD in primary care, involving dentists, pharmacists, physiotherapists, nurses and general practitioners (the UNANIME pilot study). Respir Med Res. 2021 Nov;80:100853. doi: 10.1016/j.resmer.2021.100853. Epub 2021 Aug 2. PMID 34385099